CLINICAL TRIAL: NCT04469296
Title: Trial Studying the Feasibility of a Diet Modification in pAtients With Luminal Early Breast Cancer Candidate for Primary Surgery
Brief Title: Diet Modification in pAtients With Luminal Early Breast Cancer Candidate for Primary Surgery
Acronym: MACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2019-05 MAC
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Surgery
Keywords: dietary survey,
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control arm (No Intervention): In the control arm, patients will continue their usual diet without further recommendation.
- specific diet arm "Ketogenic arm" (Experimental): In the specific diet arms, the study diet will be calculated with a dietician, for the ketogenic diet, an iso-caloric ketogenic will be proposed and explained to the patient Each diet will be respected by the patient during 9 days +/- 1 day.
  Interventions: Dietary Supplement: iso-caloric ketogenic diet
- specofoc diet arm "protein restricted diet" (Experimental): In the specific diet arms, the study diet will be calculated with a dietician, for the protein restricted diet, a 20% protein restriction as compared to the usual diet will be calculated and the diet will be explained to the patient.
  Each diet will be respected by the patient during 9 days +/- 1 day.
  Interventions: Dietary Supplement: protein restricted diet

INTERVENTIONS:
Dietary Supplement: iso-caloric ketogenic diet — Each patient will be offered a daily diet plan that includes the different groups of low glycemic index foods to bring to each meal and snack, with the notion of quantity. Carbohydrate-free foods can be consumed ad libitum. Dietary advice will be given to increase the consumption of lipid foods (vegetable oils, butter, cheeses, fatty fish, etc.) so that 65% of the total energy intake is provided by lipids. In addition, a list of unauthorized sugars and sweeteners substitutes will be proposed as well as a low glycemic index food composition table centered on carbohydrates for better control of food choice
  Arms: specific diet arm "Ketogenic arm"
Dietary Supplement: protein restricted diet — A diet reducing by 20% the amount of protein compared to the usual intake of the patient will be proposed. This new ration will be carried out by calculating the proportion of total energy intake provided by the amount of protein reduced by 20% compared to the usual intake, and by modifying lipid and carbohydrate intakes to obtain an isocaloric ration.
  Arms: specofoc diet arm "protein restricted diet"

SUMMARY:
to analyze the feasibility for patients with early luminal breast cancer to be compliant with a diet modification - ketogenic or proteins restricted diet - during 9 +/- 1 days, before breast cancer surgery.

It's a Pilot study, monocentric, randomized

DETAILED DESCRIPTION:
Many patients are modifying their diet after the diagnosis of cancer. There is a supposedly benefit, among the general public, of starving cancer cells with several diet deprivations.

Due to the lack of coherent scientific data, no evidence base recommendations can be made regarding the optimal diet during cancer and its effect on cancer growth.

The objective of this trial is to analyze the feasibility for patients with early luminal breast cancer to be compliant with a diet modification - ketogenic or proteins restricted diet - during 9 +/- 1 days, before breast cancer surgery.

The primary objective of the trial is to evaluate the compliance to the proposed diet.

The study will be conducted in patients with luminal early breast cancer, candidate to primary surgery, in order to study an homogeneous population of patients, with good performance status and without nutritional deprivation.

Metabolic changes on the main metabolic pathways and the potential antitumor effects related to these metabolic changes following the diet will be analyzed as secondary objectives of the study. We hope to find biological hypotheses to further test in a next larger prospective trial.

The impact of the patient's beliefs, anxiety and/or depression on the compliance will be analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 80 years old
* Invasive breast carcinoma, non-metastatic, stage I to III, pathologically proven, ER and/or PR positive, HER2 negative (luminal)
* No treatment yet for the current breast cancer
* Candidate for primary surgery
* Body mass index (BMI) between 18.5 and 30 for women up to 70 years old and between 21 and 30 for women between 70 and 80 years old.
* For patient ≥ 70 years, score of the Oncodage G8 questionnaire > 14 (if score ≤ 14, consultation with an oncogeriatrician required to validate the possibility of following a diet
* No addiction (alcohol, tobacco, drug, electronic cigarette) that modifies the metabolism (alcohol : ≤ 2 glasses/d or ≤10 glasses/week ; tobacco : only occasional or stopped for ≥ 6 months)
* Performance status 0-1
* Fasting blood test :

Blood cell counts : Neutrophils > 1000/µL, Platelets > 100 000/µL, Hb > 11g/dL Hepatic biology: GOT, GPT, GGT, Phosphatases alcalines < 2x normal value Renal function : clearance > 60 mL /min Lipid profile : Total cholesterol < 1.5 x normal value, HDL>0.35g/L, LDL < 2.2 g/L (<5.7 mml/L), Triglycerides < 1.5 x normal value Fasting blood glucose < 1.26 g/l Measurement of electrolytes: Potassium, Sodium, Calcium, Magnesium (according to normal laboratory values)

* ECG with a QTc interval ≤ 450 msec
* Patient able to understand, participate and give a written consent for participation to the study

Exclusion Criteria:

* Metabolic disease or other disease impairing the metabolism analysis
* High level athlete
* Unintentional weight loss ≥ 5% during the last month, or 10% during the last 6 months or compared to usual weight
* Unjustified dietary supplement (not justified by a measured deficiency) during the last month
* Restricted of unbalanced diet (vegan diet, restricted hypocaloric, hyper or hypo protein…) during the last month
* Practice of fasting during the last 3 months
* Corticoids that can't be stopped or not stopped for 2 weeks
* Mellitus diabetes (with or without insulin)
* Hypercholesterolemia requiring a treatment
* Invasive lobular carcinoma
* Pregnant or breast-feeding women
* Participation to another study with an investigational treatment during the last 30 days
* Individuals under the protection of a conservator
* Unaffiliated patient to Social Protection System.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
study of the compliance of patients to the two proposed diets. The proportion of compliant patients to the proposed diet according to the dietary survey realized during 3 days | during 3 days before the primary surgery
  A patient is considered compliant to the diet if the caloric intake is equal +/- 25% to the caloric intake of the proposed diet AND For the ketogenic diet : the carbohydrate intake is equal +/- 25% to the carbohydrate intake of the proposed diet; i.e. a carbohydrate intake between 7.5 and 12.5% of the total energy intake For the protein restricted diet, the protein intake is equal +/- 25% to the protein intake proposed for this diet; i.e. a reduction between 15 and 25% compared to the previous protein intake

SECONDARY OUTCOMES:
study of the molecular consequences of diet modifications on cancer cells and their microenvironment | At the inclusion visit and the day of surgery
  analyse markers of cell proliferation in cancer and immune cells with blood sample and tumor sample. Evaluation of markers involved in carbohydrate mitochondrial and lipid metabolism, and markers of the Pi3K-Akt-mTOR and the IGF-R pathways
study of the molecular consequences of diet modifications on cancer cells and their microenvironment | At the inclusion visit and the day of surgery
  determine the activity of the anti-tumoral immune surveillance with blood sample and tumor sample. Correlation between the cancer response and antitumoral immune with diet programm
evaluation of patient's tolerability to those diet modifications, in terms of weight status | From the inclusion visit until the Day 45 post surgery
  Weight surveillance (in kilograms)
evaluation of patient's tolerability to those diet modifications, in terms of adverse events | From the inclusion visit until the Day 45 post surgery
  monitoring of adverse events related to diet (with CTCAE (Common Terminology Criteria for Adverse Events) version 5.0)
assessment of the acceptance of study participation and reasons for refusal | During 45 days before the surgery
  Rate of patients who agreed to participate in the study compared to the total number of patients to whom the study was proposed. Collection of reasons for refusing to participate to the study
determination of the impact of diet modification on patient's quality of life | From the inclusion visit until the Day 45 post surgery
  Result of the EORTC QLQ-C30 questionnaire (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire) questionnaire
evaluation of the impact of patient's beliefs about diet and cancer on the compliance to the proposed diet. | From the inclusion visit until the Day 45 post surgery
  Result of the questionnaire of Beliefs about diet and cancer OPINELE (Opinions concernant l'alimentation, la santé et le cancer)
evaluation of the impact of the patient's anxiety and depression level on the compliance to the proposed diet | From the inclusion visit until the Day 45 post surgery
  Scores obtained on the HADS scale (Hospital Anxiety and Depression Scale) (if score or = 9, result is no significant, if sore is between 10 and 12, result is limit, if result is > or = 13, result is significant

CONTACTS AND LOCATIONS:
Overall Officials: Veronique D'HONDT, MD, Study Chair — ICM Val d'Aurelle
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all disidentified participants' data, the study protocol, the statistical analysis plan, the clinical study report and the analytic code. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Access to study data upon written detailed request sent to the institute of Montpellier Cancer (ICM), following publication and until 5 years after publication of summary data.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Result] Kushi LH, Doyle C, McCullough M, Rock CL, Demark-Wahnefried W, Bandera EV, Gapstur S, Patel AV, Andrews K, Gansler T; American Cancer Society 2010 Nutrition and Physical Activity Guidelines Advisory Committee. American Cancer Society Guidelines on nutrition and physical activity for cancer prevention: reducing the risk of cancer with healthy food choices and physical activity. CA Cancer J Clin. 2012 Jan-Feb;62(1):30-67. doi: 10.3322/caac.20140. PMID 22237782
- [Result] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Result] Cairns RA, Mak TW. Fire and water: Tumor cell adaptation to metabolic conditions. Exp Cell Res. 2017 Jul 15;356(2):204-208. doi: 10.1016/j.yexcr.2017.04.029. Epub 2017 Apr 27. PMID 28457987
- [Result] Vander Heiden MG, DeBerardinis RJ. Understanding the Intersections between Metabolism and Cancer Biology. Cell. 2017 Feb 9;168(4):657-669. doi: 10.1016/j.cell.2016.12.039. PMID 28187287
- [Result] Chen Y, Ling L, Su G, Han M, Fan X, Xun P, Xu G. Effect of Intermittent versus Chronic Calorie Restriction on Tumor Incidence: A Systematic Review and Meta-Analysis of Animal Studies. Sci Rep. 2016 Sep 22;6:33739. doi: 10.1038/srep33739. PMID 27653140
- [Result] Fontana L, Partridge L. Promoting health and longevity through diet: from model organisms to humans. Cell. 2015 Mar 26;161(1):106-118. doi: 10.1016/j.cell.2015.02.020. PMID 25815989
- [Result] Lv M, Zhu X, Wang H, Wang F, Guan W. Roles of caloric restriction, ketogenic diet and intermittent fasting during initiation, progression and metastasis of cancer in animal models: a systematic review and meta-analysis. PLoS One. 2014 Dec 11;9(12):e115147. doi: 10.1371/journal.pone.0115147. eCollection 2014. PMID 25502434
- [Result] O'Flanagan CH, Smith LA, McDonell SB, Hursting SD. When less may be more: calorie restriction and response to cancer therapy. BMC Med. 2017 May 24;15(1):106. doi: 10.1186/s12916-017-0873-x. PMID 28539118
- [Result] Weber DD, Aminzadeh-Gohari S, Tulipan J, Catalano L, Feichtinger RG, Kofler B. Ketogenic diet in the treatment of cancer - Where do we stand? Mol Metab. 2020 Mar;33:102-121. doi: 10.1016/j.molmet.2019.06.026. Epub 2019 Jul 27. PMID 31399389
- [Result] A D B. The Ketogenic Diet in Epilepsy. Can Med Assoc J. 1931 Jan;24(1):106-7. No abstract available. PMID 20318124